CLINICAL TRIAL: NCT07324278
Title: Hybrid Stroke Rehabilitation With Mirror Priming
Brief Title: Hybrid Stroke Rehab With Mirror Priming
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I-Shou University (Other)
Responsible Party: Principal Investigator, Yi-chun Li, Neuro-Rehabilitation Research Laboratory (NRRL), I-Shou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISU-OT-Li-02
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases; Stroke; Cerebrovascular Disorders
Keywords: Rehabilitation; Mirror Therapy
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose enhanced mirror priming group (Experimental)
  Interventions: Behavioral: Mirror priming; Behavioral: Conventional therapy
- Low-dose enhanced mirror priming group (Experimental)
  Interventions: Behavioral: Mirror priming; Behavioral: Conventional therapy
- Active control group (Active Comparator)
  Interventions: Behavioral: Conventional therapy

INTERVENTIONS:
Behavioral: Mirror priming — During the mirror priming process, the movement images of the participant's unaffected limb are mirrored to the affected side to provide visual feedback.
  Arms: High-dose enhanced mirror priming group; Low-dose enhanced mirror priming group
Behavioral: Conventional therapy — During conventional therapy, the participants typically receive interventions targeting the upper and lower limbs in addition to cognitive practice.

SUMMARY:
This trial aims to examine the effects of enhanced mirror priming, overcoming the limitations of traditional mirror therapy, to achieve optimization and personalized intervention.

ELIGIBILITY:
Inclusion Criteria:

1. A first-ever unilateral stroke ≥3 months
2. Age between 20 and 80 years
3. Baseline Fugl-Meyer Assessment Upper Extremity (FMA-UE) score >10
4. No severe spasticity in any joints of the affected arm
5. Ability to follow the instructions
6. No participation in other studies during the study period
7. Willingness to provide informed written consent.

Exclusion Criteria:

1. Serious medical problems or poor physical conditions that might be detrimental to study participation.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | Baseline, 2 weeks, 4 weeks, 1 month, and 3 months post-intervention.

SECONDARY OUTCOMES:
Grip and pinch power | Baseline, 4 weeks, 1 month, and 3 months post-intervention.
Revised Nottingham Sensory Assessment | Baseline, 4 weeks, 1 month, and 3 months post-intervention.
Berg Balance Scale | Baseline, 4 weeks, 1 month, and 3 months post-intervention.
Montreal Cognitive Assessment | Baseline, 4 weeks, 1 month, and 3 months post-intervention.
Motor Activity Log | Baseline, 4 weeks, 1 month, and 3 months post-intervention.
ABILHAND Questionnaire | Baseline, 4 weeks, 1 month, and 3 months post-intervention.
Chedoke Arm and Hand Activity Inventory | Baseline, 4 weeks, 1 month, and 3 months post-intervention.
Stoke Impact Scale | Baseline, 4 weeks, 1 month, and 3 months post-intervention.
Stroke Self-Efficacy Questionnaire | Baseline, 4 weeks, 1 month, and 3 months post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- E-Da Hospital, Kaohsiung City, Yanchao District, Taiwan

IPD SHARING:
Plan to Share IPD: No